CLINICAL TRIAL: NCT03956823
Title: A Cohort Study of Telmisartan on Metabolic Components and Left Ventricular Remodeling in Obese Patients With Hypertension
Brief Title: Clinical Efficacy of Telmisartan in Reducing Cardiac Remodeling Among Obese Patients With Hypertension
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: First Affiliated Hospital Xi'an Jiaotong University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: XJTU1AF-CRF-2018-005
Record Dates: First submitted 2019-05-04; First posted 2019-05-21 (Actual); Last update posted 2019-08-08 (Actual); Status verified 2019-08

CONDITIONS: Hypertension
Keywords: hypertension; obesity; telmisartan; metabolic abnormalities; cardiac remodeling
MeSH Terms: conditions — Hypertension; Obesity | interventions — Telmisartan; Amlodipine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Telmisartan (Experimental): generic name：telmisartan；dosage form：80 mg；dosage：80 mg；frequency：once a day；duration：June , 2019-June , 2021
  Interventions: Drug: telmisartan
- Amlodipine (Active Comparator): generic name： amlodipine；dosage form：5mg；dosage：5mg；frequency：once a day；duration：June , 2019-June , 2021
  Interventions: Drug: amlodipine

INTERVENTIONS:
Drug: telmisartan — Telmisartan group: telmisartan 80 mg once a day
  Arms: Telmisartan
Drug: amlodipine — amlodipine group: amlodipine 5 mg once a day
  Arms: Amlodipine

SUMMARY:
Hypertension is closely related to metabolic abnormalities such as obesity, dyslipidemia and diabetes. When hypertension is complicated with metabolic abnormalities, target organ damage is more serious, the risk of cardiovascular adverse events is greater, and the treatment is more complex. The pathophysiological mechanism of obesity-associated hypertension has its particularity. Blood pressure control and effective control of obesity are important therapeutic targets. At present, there are no guidelines for the treatment of obesity-associated hypertension. Although several drugs have certain effects on fat metabolism, they have little effect on blood pressure and have some side effects in long-term use. Among the existing antihypertensive drugs, angiotensin II type 1 receptor (AT-1) antagonists have shown their particularity in improving glycolipid metabolism, but strict clinical trials are needed to confirm their effectiveness in weight loss and metabolism improvement. Previous studies have shown that obese patients with hypertension have severe insulin resistance, poor glycolipid metabolism and are prone to cardiovascular damage. Telmisartan can block AT-1 receptor and partially activate PPAR-γ, increase the expression of PPAR-γ target gene in preadipocytes, improve the function of visceral adipose tissue, and effectively prevent obesity-related cardiovascular diseases. It is presumed that telmisartan can act as a PPAR-γ agonist in clinic by altering the metabolic components and insulin sensitivity, but there is no clinical evidence for this. On the basis of previous studies, this study aims to evaluate the clinical efficacy of telmisartan or amlodipine in controlling blood pressure, reducing fat accumulation, improving insulin sensitivity, and reducing cardiac remodeling in obese patients with hypertension by prospective cohort study.

DETAILED DESCRIPTION:
At present, there are no guidelines for the treatment of obese patients with hypertension. Blood pressure control and effective control of obesity are important therapeutic targets for obesity-associated hypertension. Whether telmisartan can be used as PPAR-γ agonist, unlike other AT-1 receptor antagonists and calcium channel blockers amlodipine, can improve the visceral adipose tissue function and cardiac remodeling in obese patients with hypertension by altering their metabolic components and insulin sensitivity while controlling blood pressure. There is no evidence that telmisartan can reduce cardiac remodeling in obese patients with hypertension.

1.Research contents:

1. To evaluate the clinical efficacy of telmisartan or amlodipine in controlling blood pressure, reducing fat accumulation, improving glycolipid metabolism and insulin sensitivity, and reducing cardiac remodeling in obese patients with hypertension;
2. To evaluate whether telmisartan can alter metabolic components and insulin sensitivity, improve visceral adipose tissue function and reduce cardiac remodeling in obese patients with hypertension by blocking AT-1 receptor and partially activating PPAR-gamma, which is different from other AT-1 receptor antagonists and calcium channel blockers amlodipine.

2.Research population 2.1 Entry criteria

Only those who possess the following four conditions can enter the study:

1. Essential hypertension patients (including confirmed hypertension without regular treatment, average blood pressure (≥160 or/and 100 mmHg) in two follow-up visits; or hypertension under combined antihypertensive treatment; or unsatisfactory blood pressure control with single drug treatment, blood pressure above 140 or/and 90 mmHg)；
2. Age ranges from 18 to 79；
3. Body mass index, BMI (≥30 kg/m2), or waist circumference, male (≥102 cm), female (≥ 88 cm)；
4. Ability to provide informed consent。

2.2 exclusion criteria

One of the following is not included:

(1) secondary hypertension; (2) acute cardiovascular and cerebrovascular events within 3 months; (3) severe cardiomyopathy, rheumatic heart disease, congenital heart disease;(4) unstable angina pectoris; (5) severe liver or kidney disease (ALT increased by 2 times; Creatinine > 2. 5 mg/dL); (6) malignant tumors; (7) gout; (8) women who are taking birth control pills or are at risk of pregnancy; (9) have a history of allergy to research drugs; (10) patients with specific contraindications to the study drugs; (11) participants in other clinical trials; (12) patients with difficulty in long-term follow-up or poor compliance; (13) the competent doctor considers it inappropriate to participate in clinical research.

3.The input information of the subjects

1. Sample source: Since December 2018, patients with essential hypertension were diagnosed in the First Affiliated Hospital of Xi'an Jiaotong University and treated with telmisartan or amlodipine alone under the guidance of doctors；
2. Recruitment procedures: selecting the subjects according to inclusion and exclusion criteria, and signing informed consent.

4.Criteria for termination or withdrawal of research subjects

1. Those who need revascularization because of myocardial infarction and unstable angina pectoris;
2. Heart failure;
3. Stroke.

5. Study Groups

1. Telmisartan group: Telmisartan 80 mg once a day
2. amlodipine group: amlodipine 5 mg once a day

6.Research evaluation index

1. Baseline indicators: age, sex, occupation, height, weight, BMI, waist-hip circumference, systolic blood pressure, diastolic blood pressure, heart rate;
2. Metabolic indicators: blood lipid, liver function, kidney function, oral glucose tolerance test, simultaneous insulin release test, plasma Glucagon, plasma aldosterone, plasma angiotensin II, abdominal fat distribution
3. Fat function: serum leptin, serum adiponectin, serum TNFalpha, serum IL-6, serum hs-CRP, serum PPAR-γ;
4. Cardiac remodeling: echocardiographic parameters .

7.Research steps

1. Clinical trials are ethically reviewed by ethics committees, and clinical trials are registered;
2. Collect cases according to inclusion and exclusion criteria, collect medical history data of subjects, and complete follow-up. At the same time, clinical and biochemical experiments were carried out;
3. Comprehensive analysis of experimental data, repetition and supplementation of necessary molecular biological experiments, comprehensive summary of the results, writing and publishing SCI papers and Chinese core journal papers.

ELIGIBILITY:
Inclusion Criteria:

* Essential hypertension patients (including those with unconventional diagnosed hypertension, whose average blood pressure was more than 160 or/and 100 mmHg in two outpatient follow-up visits; or those who were undergoing combined antihypertensive therapy; or those whose blood pressure control was unsatisfactory and whose blood pressure was more than 140 or/and 90 mmHg in single drug treatment);
* The age ranged from 18 to 79 years;
* Body mass index, BMI (≥ 30 kg/m2), or waist circumference, male (≥102 cm), female (≥88 cm);
* Ability to provide informed consent.

Exclusion Criteria:

* Secondary hypertension;
* Acute cardiovascular and cerebrovascular events occurred within 3 months;
* Complicated with severe cardiomyopathy, rheumatic heart disease, congenital heart disease;
* unstable angina pectoris;
* Severe liver or kidney diseases (ALT increased twice; creatinine > 2.5 mg/d1);
* Tumor；
* Gout;
* Women who are taking contraceptives or are at risk of pregnancy; -Has a history of allergy to research drugs;
* Those who have clear contraindications to the research drugs;
* Those who are participating in other clinical trials;
* Those who are not easy to follow up for a long time or have poor compliance;
* Doctors in charge do not consider it advisable to participate in clinical research.

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2019-08-01 (Actual); Primary Completion 2021-05-01 (Estimated); Study Completion 2021-12-01 (Estimated)

PRIMARY OUTCOMES:
Revascularization for myocardial infarction and unstable angina pectoris | From date of randomization until the date of first documented progression，assessed up to 24 months
  Revascularization for myocardial infarction and unstable angina pectoris
Heart failure | From date of randomization until the date of first documented progression，assessed up to 24 months
  Heart failure
stroke | From date of randomization until the date of first documented progression，assessed up to 24 months
  stroke

CONTACTS AND LOCATIONS:
Overall Officials: Gang Tian, doctor, Principal Investigator — First Affiliated Hospital Xi'an Jiaotong University
Locations (1):
- First Affiliated Hospital of Xi'an Jiaotong University, Xi’an, Shanxi, China

IPD SHARING:
Plan to Share IPD: No